CLINICAL TRIAL: NCT02300168
Title: Neuromuscular Blockade as a Determinant of Surgical Outcome and Post-operative Recovery, in Patients Undergoing Elective Laparoscopic Bariatric Surgery
Brief Title: Neuromuscular Blockade: Outcome and Recovery for Laparoscopic Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Pierre Garneau, Chief, General Surgery Department, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Other Study IDs: MISP-51834
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Bariatric Surgery Candidate
Keywords: bariatric surgery; neuromuscular blockade

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Laparoscopic sleeve gastrectomy (LSG) is a restrictive procedure which consists in creating a narrow tube-like stomach, designed to decrease appetite by reducing the ability of the stomach to distend.

SUMMARY:
The aim of the current observational study is to better assess the relationships between neuromuscular blockade and multiple surgical outcomes in patients undergoing elective laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
Performing bariatric surgery as a short-stay procedure is an ongoing trend in many centers around the world. For morbidly obese (MO) patients, the anesthetic approach is based on choosing drugs that have the least potential for accumulation. This allows a more rapid and clear-headed recovery and contributes to reduced duration of perioperative time. However, when neuromuscular blockade (NMB) is required during surgery, complete recovery is a major factor that may prevent from a rapid fast-track discharge.

In Canada, reversal of NMB is achieved by using acetylcholinesterase (AChE) inhibitors, mostly neostigmine, which must be administered after a certain level of spontaneous recovery in order to ensure a complete reversal. This elongates the time spent in the operating room (OR), and prevent therefore from a fast track surgery procedure. On the other hand, in an effort to shorten the time spent in the OR, AChE inhibitors may sometime be administered too early before spontaneous recovery, and post-operative residual curarization (PORC) may then be observed. In the post-anesthesia care unit (PACU), PORC may be particularly problematic, because of the possible occurrence of critical respiratory events (CREs). This in turn is also associated with significant delayed discharges.

Because of the aforementioned inconveniences, Canadian anesthesiologists are reluctant to induce deep NMB. Consequently, intra-abdominal pressure remain non optimal during the surgery, which do not facilitate the surgeons work, in addition to increase perioperative time. This problem is particularly frequent in cases of bariatric surgeries.

The current study will explore this question from the perspective of the surgeon satisfaction and the patient quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

MO patients [body mass index (BMI)≤ 55kg/m2] scheduled for elective laparoscopic sleeve gastrectomy under general anesthesia.

Exclusion Criteria:

* a physical status >3 (ASA),
* a difficult tracheal intubation,
* a known or suspected disorder affecting NMB,
* a renal, pulmonary, cardiac, and/or hepatic dysfunction,
* malignant hyperthermia,
* pregnancy, breastfeeding,
* allergy or contraindication to narcotics, rocuronium, neostigmine, or other medications used during anesthesia
* patients with sleep apnea syndrome will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MO patients from the bariatric surgery department of Hopital Sacre Coeur de Montreal
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
surgeon evaluation of working surgical conditions | intraoperative
  the surgeon will score the surgical working conditions at 15 min intervals, according to a 5-point ordinal scale

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Y Garneau, MD, Principal Investigator — Hopital Sacre Coeur de Montreal

REFERENCES:
- [Result] Raeder J. Bariatric procedures as day/short stay surgery: is it possible and reasonable? Curr Opin Anaesthesiol. 2007 Dec;20(6):508-12. doi: 10.1097/ACO.0b013e3282f09443. PMID 17989541
- [Result] Servin F. Ambulatory anesthesia for the obese patient. Curr Opin Anaesthesiol. 2006 Dec;19(6):597-9. doi: 10.1097/ACO.0b013e328010cb78. PMID 17093361
- [Result] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- [Result] Butterly A, Bittner EA, George E, Sandberg WS, Eikermann M, Schmidt U. Postoperative residual curarization from intermediate-acting neuromuscular blocking agents delays recovery room discharge. Br J Anaesth. 2010 Sep;105(3):304-9. doi: 10.1093/bja/aeq157. Epub 2010 Jun 24. PMID 20576632